CLINICAL TRIAL: NCT03872284
Title: Study of Neuro-ophthalmology Disorders in Autoimmune Encephalitis (NODE)
Brief Title: Neuro-ophthalmology and Autoimmune Encephalitis (NODE)
Acronym: NODE
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0749; 2019-A00684-53 (Other: ID RDB)
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Autoimmune Encephalitis
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 1: Patients in the study group have a diagnosis of autoimmune encephalitis, are 18 to 70 years old, and have no significant comorbidity such as psychiatric, neurological conditions and able to understand the aim of this study.
  Interventions: Other: oculomotor movement recordings, neurovisual assessment

INTERVENTIONS:
Other: oculomotor movement recordings, neurovisual assessment — Each participant will have a neurovisual assessment and an oculomotor movement recording with an eye tracker (infra red cameras).

SUMMARY:
Autoimmune encephalitis represents a group of rare and heterogeneous neurological disorders. Pathophysiological mechanisms in these diseases are still unknown. Recently, oculomotor and neurovisual disorders have been described. Cerebral areas and neuronal networks associated with these abnormalities are well described. The investigator proposes to study and describe such neuro-ophthalmological disorders in a prospective cohort of patients with a autoimmune encephalitis, to better understand the pathophysiological basis of this neurological condition.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of autoimmune encephalitis
* With or without pathological antibody
* Aged from 18 to 70 years old
* Able to understand the aims and methods of this project
* Non opposed to the participation of this study

Exclusion Criteria:

* Other neurological, psychiatric or systemic conditions, which could induce neuro-ophthalmological signs Cognitive impairment, which is not linked to autoimmune encephalitis
* Ophthalmological condition, which could modify the interpretation of neuro-ophthalmological data Inability to remain seated
* Pregnancy or breast feeding
* Adults under guardianship

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women 18 to 70 years old diagnosed with autoimmune encephalitis
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
Percentage of patients presenting a neuro-ophthalmological abnormality. | Day 0
  A neuro-ophthalmological disorder is defined as an abnormality in the oculo-motor movement recording or/and the presence of a neurovisual impairment.
Percentage of patients presenting neuro-ophthalmological abnormality. | At 6 months if an abnormality is found
  A neuro-ophthalmological disorder is defined as an abnormality in the oculo-motor movement recording or/and the presence of a neurovisual impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Tilikete, Prof., Principal Investigator — Department of neuro-ophthalmology, Pierre Wertheimer university hospital
Locations (1):
- Hospices Civils de Lyon, Bron, France